CLINICAL TRIAL: NCT06694558
Title: Monocytes in Subjects With Type 1 Diabetes and Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Stanford University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-1015; K12DK133995 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease(CKD); Type 1 Diabetes (T1D)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Type 1 Diabetes: Patients with Type 1 Diabetes with or without chronic kidney disease

SUMMARY:
This is a cross-sectional study in patients with Type 1 diabetes (TID) and chronic kidney disease (CKD) to test if time in range (TIR) affects the degree of hyperglycemia required for monocyte activation, podocyte injury, and assess if monocyte activation is attenuated by glucagon-like peptide (GLP-1) agonist treatment ex vivo.

DETAILED DESCRIPTION:
The monocyte response from patients with T1D CKD will be compared to monocytes from T1D subjects without CKD as a control. Potential subjects will be recruited from existing Cleveland Clinic patients or the community. The study will entail an initial phone screen followed by a formal screening visit to determine eligibility. Eligible subjects will return for a study visit within 4 weeks for a blood draw. There is no intervention. This will complete the study for subjects unless the investigators do not obtain enough monocytes from the initial blood draw to complete the requisite lab studies. If this occurs, the investigators will ask the patient to return for a repeat study visit. All endpoints evaluating monocyte and podocyte injury will be conducted in the lab ex vivo.

ELIGIBILITY:
Inclusion Criteria:

1. T1D CKD subjects:

   1. Adults, males or females diagnosed with T1D
   2. Age 18-65 years
   3. Diagnosed with CKD (eGFR 60-90 ml/min/1.73 m2)
   4. Diagnosed with albuminuria (UACR 30-500 mg/g)
   5. On insulin injections or pump
   6. On CGM

   Based on baseline CGM metrics, the investigators will stratify subjects to 2 groups Group A (Lower TIR group): TIR<60%, A1c 7.5-9.5 Group B (Higher TIR group): TIR>70% A1c 5.0-7.0
2. Controls: T1D subjects without CKD

   1. Adults, males or females diagnosed with T1D
   2. Age 18-65 years
   3. No CKD (eGFR >90 ml/min/1.73 m2)
   4. No albuminuria (UACR <30 mg/g)
   5. On insulin injections or pump
   6. On CGM

Based on baseline CGM metrics, the investigators will stratify subjects to 2 groups Group A (Lower TIR group): TIR<60%, A1c 7.5-9.5 Group B (Higher TIR group): TIR>70% A1c 5.0-7.0

Exclusion Criteria:

1. Hemoglobin <9
2. On GLP-1 agonist or DPP4 inhibitor or sodium-glucose co-transporter-2 inhibitors use within 30 days
3. pregnancy or plans to become pregnant
4. On steroids
5. Diagnosed with cancer, immunosuppression/autoimmune conditions
6. Reported heavy alcohol use or recreational drug use
7. Any condition which jeopardizes patient safety or affects monocytes at physician's discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 1 Diabetes with or without chronic kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with proinflammatory monocytes by flow cytometry, higher ER stress, and cytokine levels after monocyte exposure to hyperglycemia compared to euglycemia for 6 hours. | monocyte response to varying glycemic exposure after 6 hrs
  Number of subjects with proinflammatory monocytes by flow cytometry, higher ER stress, and cytokine levels after monocyte exposure to hyperglycemia compared to euglycemia for 6 hours

SECONDARY OUTCOMES:
Number of subjects with monocytes which induces higher podocyte injury after monocyte exposure to hyperglycemia compared to euglycemia for 6 hours. | monocyte response to varying glycemic exposure after 6 hrs
  Number of subjects with monocytes which induces higher podocyte injury after monocyte exposure to hyperglycemia compared to euglycemia for 6

CONTACTS AND LOCATIONS:
Overall Officials: Rong M Zhang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT06694558/Prot_SAP_000.pdf